CLINICAL TRIAL: NCT06158191
Title: Abdominal Obesity as a Therapeutic Target: Long-term Benefits of Abdominal Fat Loss and Weight Stabilization in High-risk Abdominally Obese Dyslipidemic Patients With the Features of the Metabolic Syndrome (SYNERGIE Study)
Brief Title: Long-term Benefits of Abdominal Fat Loss in Abdominally Obese Dyslipidemic Patients (SYNERGIE Study)
Acronym: SYNERGIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Pierre DESPRÉS, PhD, Principal Investigator, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYNERGIE Study
Record Dates: First submitted 2023-11-14; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Obesity, Visceral; Diet, Healthy; Cardiometabolic Syndrome; Lifestyle-related Condition
Keywords: Cardiometabolic health; Physical activity; Diet; Visceral obesity; Lifestyle intervention; Cardiorespiratory fitness
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome; Mental Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention group and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Lifestyle modification program focused on physical activity and diet. Diet recommendations in line with the AHA's guidelines focusing on foods rather than nutrients. Emphasis will be placed on awareness of the risk of overeating associated with the consumption of energy-dense foods (fat, added sugar or both). Dieticians will closely interact with participants and will not recommend a daily energy deficit greater than 500 kcal. Participants will have constant access to the dieticians and bi-monthly appointment will be required for the first year of the study to tailor recommendations to the participants. The physical activity/exercise component will be under the supervision of a kinesiologist and will aim at 160 minutes per week of moderate intensity endurance-exercise (mainly brisk walking) tailored to the participants' preferences and habits. Following the first year, participants will meet a dietician and a kinesiologist every month for the next two years (maintenance period).
  Interventions: Behavioral: Lifestyle modification program
- Control group (No Intervention): Usual behavior

INTERVENTIONS:
Behavioral: Lifestyle modification program — Participants will take part in a lifestyle modification program focused on physical activity and diet.
  Arms: Intervention group

SUMMARY:
The objective of this clinical trial is to verify whether the beneficial effects of weight loss on visceral fat measured by computed tomography and metabolic risk factors for coronary heart disease are maintained once high-risk patients without symptoms and with visceral obesity and dyslipidemia are stabilized and maintained for two additional years after a one-year weight loss (5-10%) program.

Before entering the study, after the one-year intervention program, and after the 2-year maintenance period, participants will be asked to take part in multiple assessments: fasting lipid profile and apolipoproteins measurements, oral glucose tolerance test, anthropometric measurements, computed tomography, dual-energy X-ray absorptiometry, oral lipid tolerance test, measurements of inflammatory markers, physical activity and dietary diaries, cardiorespiratory fitness assessed by a submaximal treadmill test, and measurements of resting and exercise blood pressure.

During the one-year intervention, participants will be closely monitored by the study's dietitians and kinesiologists to achieve the target weight loss. Dieticians will not recommend a daily energy deficit greater than 500 calories and will focus on foods rather than the nutrient composition of the diet. Participants will have access to the dieticians at all time, and appointments every two months will be required during the first year. Regarding physical activity, kinesiologists will supervise the exercise prescription which will aim at 160 minutes per week of moderate-intensity aerobic-exercise. The physical activity prescription will be adjusted by the kinesiologist according to the participant's preferences and habits.

The investigators hypothesize that there will be a worsening in some features of the metabolic syndrome over the two-year weight maintenance period. However, it is suggested the greater the weight loss during the intervention, the less marked the deterioration will be. Finally, the investigators put forward that even in the absence of weight loss during the intervention, the lifestyle modification program will prevent visceral fat accumulation expected to be observed over the two-year maintenance period in the control group maintaining their usual behaviour.

DETAILED DESCRIPTION:
Because of the risk of chronic complications associated with this condition, obesity has become a source of concern for health authorities of countries confronted to the consequences of the affluent and sedentary lifestyle of most of their citizens. It is also finally acknowledged that there is a need to go beyond the study of biological factors promoting obesity and to document approaches, both at the individual and society levels, likely to have an impact on the adiposity of the population of all ages and on related indicators of health and well-being.

In this context, the principal investigator's laboratory has ben studying the metabolic complications of obesity for over thirty years, with a major focus on adipose tissue, lipid metabolism and cardiovascular disease risk factors. It has been particularly involved in studies investigating the seemingly paradoxical and puzzling metabolic heterogeneity of obesity. Imaging studies conducted in the investigator's laboratory have shown that, in both men and women and irrespective of the variation in the amount of total body fat, patients with visceral obesity are characterized by the most severe metabolic abnormalities. Despite these findings, no study has shown that aiming at visceral adipose tissue loss as a therapeutic target would reduce the risk of coronary heart disease (CHD) in patients characterized by this condition. The best available data on the long-term benefits of moderate weight loss come from two landmark trials: the Finnish Prevention of Diabetes study and the American Prevention Program. Despite these trials providing evidence that moderate weight loss produced by an improved diet and a more physically active lifestyle can decrease the risk of developing type 2 diabetes in a high-risk population, several questions remain unanswered. Was the substantial reduction in risk of developing diabetes related to a selective loss of visceral adipose tissue? Was the assumed loss of visceral adipose tissue maintained throughout the two trials? Is the loss of visceral adipose tissue induced by moderate weight loss maintained once a reduced body weight is achieved and maintained over time? Would the assumed improvements in metabolic risk factors produced by these lifestyle modification programs be sustained had the reduced body weight been maintained over time? Most studies have assessed the potential metabolic benefits of weight loss immediately at the end of the weight loss intervention program. Although precautions have often been taken to perform this metabolic assessment once body weight is stabilized (and therefore when patients are presumably in energy balance), whether such improvements in the features of the metabolic syndrome would be maintained over time had patients been able to successfully maintain their reduced body weight over months, if not years, remains unclear. Therefore, there is an urgent need to properly document not only changes in the features of the metabolic syndrome in response to losses of abdominal fat and of total body fat, but also to verify whether the expected metabolic benefits are maintained over time if patients successfully maintain their recommended moderate (5-10%) weight reduction. The investigators consider that this therapeutic objective is realistic and achievable, but the notion that it is enough to generate a sustained and substantial improvement in all markers of the metabolic syndrome modulating CHD risk need to be secured. They hypothesized that under conditions of weight maintenance at a reduced body weight (between 5-10%), there will be a differential deterioration in some features of the metabolic syndrome over the two-year weight maintenance period. However, the investigators propose that such deterioration will be less marked when body weight is reduced by closer to 10% of the initial body weight and maintained as compared to lesser reductions. Finally, the investigators put forward the hypothesis that even in the absence of weight loss, the lifestyle intervention program will prevent visceral adipose tissue accumulation expected to be observed over the two-year follow-up period in the control group maintaining their usual behaviour.

These hypotheses have never been tested, particularly in the population of high-risk viscerally obese patients with the proper measurement of relevant features of the metabolic syndrome. In addition, whether physical activity and an improved diet could have an impact on visceral adipose tissue loss and related metabolic complications even in the absence of weight loss is a question of considerable clinical importance that is still a matter of debate and requires further evidence.

The overall objective of this trial is to verify whether the beneficial effects of weight loss on visceral adipose tissue measured by computed tomography and metabolic risk factors for CHD are maintained once asymptomatic but high-risk patients with abdominal obesity and hypertriglyceridemia are stabilized and maintained for two additional years after a one-year weight loss (5-10%) program. The secondary objectives of the study include:

To document the magnitude of changes of a comprehensive set of atherogenic-prothrombotic-inflammatory risk markers including postprandial lipemia in response to a 5-10% weight loss produced over a period of one year in a sample of asymptomatic but high-risk men with visceral obesity and hypertriglyceridemia.

To compare the differential response of metabolic risk factors (including potential changes in visceral adipose tissue) during the two-year weight maintenance phase after a 5-10% reduction in body weight.

To document the potential deterioration in a comprehensive set of metabolic risk variables in a group of asymptomatic but high-risk men with visceral obesity and hypertriglyceridemia maintaining their usual behaviour (control group).

To document the long-term effects of a lifestyle modification program not inducing weight loss (non-responders of the lifestyle modification program) on a comprehensive set of metabolic risk variables (including visceral adipose tissue) in asymptomatic but high-risk men with visceral obesity and hypertriglyceridemia.

Among patients achieving a 5-10% weight loss over the first year of the study, to quantify the proportion of men who will be able to maintain such a reduced body weight over an additional period of two years if offered close counselling and monitoring by a team of health professionals.

For this study, 186 asymptomatic high-risk men with features of the metabolic syndrome will be assigned to either:

a control group (n=42) receiving a medical, morphometric and metabolic evaluation at baseline as well as usual diet and physical activity recommendations (maintaining their usual behaviour) with follow-up measurements at years 1, 2 and 3;

another group (n=144) subjected to the same baseline and follow-up measurements but who would benefit from a monthly individualized dietary counselling combined with a supervised exercise/physical activity program expected to generate a 5-10% weight loss over a period of one year.

After the first year, the recommendations provided by the study dieticians and kinesiologist will be adjusted to aim at the maintenance of body weight for two additional years. Although the objective of the present study is to reshape the lifestyle of sedentary participants with abdominal obesity so that significant weight loss is achieved over a year, it is expected that some subjects will show a rebound of their body weight during the two-year weight maintenance period. These subjects will be kept in the program for ethical reasons, but two sets of analyses will be conducted at the end of the study: 1- analyses on subjects that have been able to maintain their body weight during the weight maintenance phase within a variation below 2.5% and 2- analyses on all subjects on an intent-to-treat basis.

The investigators expect a 5-10% weight loss to induce a 20-40% loss of visceral adipose tissue. The present study has been powered (80% power) to detect a difference of 20% in changes in visceral adipose tissue as statistically significant. Two statistical approaches will be conducted to analyze data. First, a two-way analysis of variance will be used to analyze data at baseline and at one year; one experimental factor being the comparison among the two groups (the fixed factor being the various interventions) whereas the other being the testing phase (baseline and one year). Time will be analyzed as a repeated-measure factor. Different statistical models will be used to obtain the best-fit model and likelihood ratio tests will be carried out between models contained in the others. Comparisons of Akaike's information criterion (AIC) for the different models will also be performed. Normality will be verified with Shapiro-Wilk and Mardia tests. The second approach to analyze the data will be similar to the first one except for the definition of the factor time which will have in this case three levels: year 1, year 2 and year 3. Values at baseline will be used as covariates. This approach will allow us to test the possibility that the non responders were different at baseline from other participants assigned in the weight loss group. In addition, canonical analysis will be performed to identify relationships between two sets of variables to find the linear combination of adiposity variables (BMI, fat mass, subcutaneous and visceral adipose tissue) that will be most significantly correlated with the linear combination of metabolic risk factors. Posteriori comparisons between means will be obtained using Tukey's technique. Significance will be set at p-values ≤ 0.05. Analyses will be conducted using SAS (SAS Institute Inc, Cary, NC, USA) under the guidance of the research center's statistician.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 25 kilograms/meters² and 40 kilograms/meters²
* Waist circumference ≥ 90 centimeters and triglycerides ≥ 2.0 milimoles/liter or HDL < 1.03 milimoles/liter

Exclusion Criteria:

* Pharmacological treatment for hypertension, dyslipidemias, type 2 diabetes, coronary heart disease, or cardiovascular disease
* Type 2 diabetes diagnosis at baseline screening
* Use of weight loss medication in the past 6 months

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2004-03-26 (Actual); Primary Completion 2008-12-15 (Actual); Study Completion 2008-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in body weight following the lifestyle intervention and the maintenance period using dual-energy x-ray absorptiometry | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in body weight in kilograms
Changes in visceral adipose tissue area following the lifestyle intervention and the maintenance period using computed tomography | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in visceral adipose tissue area in centimeters²
Changes in visceral adipose tissue volume following the lifestyle intervention and the maintenance period using computed tomography | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in visceral adipose tissue volume in centimeters³
Changes in waist circumference following the lifestyle intervention and the maintenance period using a standardized measuring tape | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in waist circumference in centimeters
Changes in subcutaneous adipose tissue area following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in subcutaneous adipose tissue area in centimeters²
Changes in subcutaneous adipose tissue volume following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in subcutaneous adipose tissue volume in centimeters³

SECONDARY OUTCOMES:
Changes in systolic blood pressure following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in systolic blood pressure in mercury millimeters
Changes in diastolic blood pressure following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in diastolic blood pressure in mercury millimeters
Changes in plasma triglycerides following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in plasma triglycerides in millimoles per liter
Changes in fasting total cholesterol following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fasting total cholesterol in millimoles per liter
Changes in fasting HDL cholesterol following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fasting HDL cholesterol in millimoles per liter
Changes in fasting LDL cholesterol following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fasting LDL cholesterol in millimoles per liter
Changes in fasting apolipoproteinA1 following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fasting ApolipoproteinA1 in grams per liter
Changes in fasting apolipoproteinB following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fasting ApolipoproteinB in grams per liter
Changes in fasting glucose following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fasting glucose in millimoles per liter
Changes in fasting insulin following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fasting insulin in picomoles per liter
Changes in glucose area under the curve after an oral glucose tolerance test following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in glucose area under the curve in millimoles per liter * 180 minutes
Changes in insulin area under the curve after an oral glucose tolerance test following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in insulin area under the curve in picomoles per liter * 180 minutes
Changes in insulin resistance following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in insulin resistance assessed by the homeostasis model assessment of insulin resistance (HOMA-IR)
Changes in cardiorespiratory fitness following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in Metabolic Equivalent of Tasks (METs) reach at a heart rate of 150 beats per minutes
Changes in physical activity behaviours following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in daily physical activity practice according to the three-day Bouchard physical activity journal. Days in the journal were divided into 15-min periods and energy expenditure was qualified on a scale of 1 to 9 for each period. A higher number indicates a greater energy expenditure for that period.
Changes in the number of steps per day following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in the number of steps per day with a pedometer
Changes in total energy intake following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in total energy intake in kilocalories
Changes in the macronutrient composition of the diet following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in the macronutrient composition of the diet in percentage
Changes in fat mass following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fat mass in kilograms
Changes in fat-free mass following the lifestyle intervention and the maintenance period | After the 1-year intervention and at 3 years after the beginning of the study
  Changes in fat-free mass in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Després, Ph.D., Principal Investigator — Laval University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrett-Connor EL. Obesity, atherosclerosis, and coronary artery disease. Ann Intern Med. 1985 Dec;103(6 ( Pt 2)):1010-9. doi: 10.7326/0003-4819-103-6-1010. PMID 3904565
- [Background] Bray G, Bouchard C, James W. Handbook of obesity. United States of America: Marcel Dekker, Inc.; 1998
- [Background] Hubert HB, Feinleib M, McNamara PM, Castelli WP. Obesity as an independent risk factor for cardiovascular disease: a 26-year follow-up of participants in the Framingham Heart Study. Circulation. 1983 May;67(5):968-77. doi: 10.1161/01.cir.67.5.968. PMID 6219830
- [Background] Kissebah AH, Freedman DS, Peiris AN. Health risks of obesity. Med Clin North Am. 1989 Jan;73(1):111-38. doi: 10.1016/s0025-7125(16)30695-2. PMID 2643000
- [Background] Manson JE, Colditz GA, Stampfer MJ, Willett WC, Rosner B, Monson RR, Speizer FE, Hennekens CH. A prospective study of obesity and risk of coronary heart disease in women. N Engl J Med. 1990 Mar 29;322(13):882-9. doi: 10.1056/NEJM199003293221303. PMID 2314422
- [Background] National Institutes of Health. The practical guide. Identification, evaluation, and treatment of overweight and obesity in adults. National Heart, Lung, and Blood Institute and North American Association for the Study of Obesity; October 2000:1-77
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Despres JP. The insulin resistance-dyslipidemia syndrome: the most prevalent cause of coronary artery disease? CMAJ. 1993 Apr 15;148(8):1339-40. No abstract available. PMID 8462056
- [Background] Després JP. Visceral obesity: A component of the insulin resistance-dyslipidemic syndrome. Can J Cardiol. 1994;10:17B-22B.
- [Background] Després JP. Obesity and lipid metabolism: relevance of body fat distribution. Curr Opin Lipidol. 1991;2:5-15.
- [Background] Despres JP. Lipoprotein metabolism in visceral obesity. Int J Obes. 1991 Sep;15 Suppl 2:45-52. No abstract available. PMID 1794938
- [Background] Despres JP, Couillard C, Gagnon J, Bergeron J, Leon AS, Rao DC, Skinner JS, Wilmore JH, Bouchard C. Race, visceral adipose tissue, plasma lipids, and lipoprotein lipase activity in men and women: the Health, Risk Factors, Exercise Training, and Genetics (HERITAGE) family study. Arterioscler Thromb Vasc Biol. 2000 Aug;20(8):1932-8. doi: 10.1161/01.atv.20.8.1932. PMID 10938014
- [Background] Despres JP, Moorjani S, Ferland M, Tremblay A, Lupien PJ, Nadeau A, Pinault S, Theriault G, Bouchard C. Adipose tissue distribution and plasma lipoprotein levels in obese women. Importance of intra-abdominal fat. Arteriosclerosis. 1989 Mar-Apr;9(2):203-10. doi: 10.1161/01.atv.9.2.203. PMID 2923576
- [Background] Despres JP, Nadeau A, Tremblay A, Ferland M, Moorjani S, Lupien PJ, Theriault G, Pinault S, Bouchard C. Role of deep abdominal fat in the association between regional adipose tissue distribution and glucose tolerance in obese women. Diabetes. 1989 Mar;38(3):304-9. doi: 10.2337/diab.38.3.304. PMID 2645187
- [Background] Lemieux S, Despres JP. Metabolic complications of visceral obesity: contribution to the aetiology of type 2 diabetes and implications for prevention and treatment. Diabete Metab. 1994 Jul-Aug;20(4):375-93. No abstract available. PMID 7843469
- [Background] Lemieux S, Despres JP, Moorjani S, Nadeau A, Theriault G, Prud'homme D, Tremblay A, Bouchard C, Lupien PJ. Are gender differences in cardiovascular disease risk factors explained by the level of visceral adipose tissue? Diabetologia. 1994 Aug;37(8):757-64. doi: 10.1007/BF00404332. PMID 7988777
- [Background] Pascot A, Lemieux I, Prud'homme D, Tremblay A, Nadeau A, Couillard C, Bergeron J, Lamarche B, Despres JP. Reduced HDL particle size as an additional feature of the atherogenic dyslipidemia of abdominal obesity. J Lipid Res. 2001 Dec;42(12):2007-14. PMID 11734573
- [Background] Pouliot MC, Despres JP, Nadeau A, Moorjani S, Prud'Homme D, Lupien PJ, Tremblay A, Bouchard C. Visceral obesity in men. Associations with glucose tolerance, plasma insulin, and lipoprotein levels. Diabetes. 1992 Jul;41(7):826-34. doi: 10.2337/diab.41.7.826. PMID 1612197
- [Background] Tchernof A, Lamarche B, Prud'Homme D, Nadeau A, Moorjani S, Labrie F, Lupien PJ, Despres JP. The dense LDL phenotype. Association with plasma lipoprotein levels, visceral obesity, and hyperinsulinemia in men. Diabetes Care. 1996 Jun;19(6):629-37. doi: 10.2337/diacare.19.6.629. PMID 8725863
- [Background] Couillard C, Bergeron N, Prud'homme D, Bergeron J, Tremblay A, Bouchard C, Mauriege P, Despres JP. Postprandial triglyceride response in visceral obesity in men. Diabetes. 1998 Jun;47(6):953-60. doi: 10.2337/diabetes.47.6.953. PMID 9604874
- [Background] Tchernof A, Labrie F, Belanger A, Prud'homme D, Bouchard C, Tremblay A, Nadeau A, Despres JP. Androstane-3alpha,17beta-diol glucuronide as a steroid correlate of visceral obesity in men. J Clin Endocrinol Metab. 1997 May;82(5):1528-34. doi: 10.1210/jcem.82.5.3924. PMID 9141545
- [Background] Lemieux I, Pascot A, Prud'homme D, Almeras N, Bogaty P, Nadeau A, Bergeron J, Despres JP. Elevated C-reactive protein: another component of the atherothrombotic profile of abdominal obesity. Arterioscler Thromb Vasc Biol. 2001 Jun;21(6):961-7. doi: 10.1161/01.atv.21.6.961. PMID 11397704
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Doucet E, Imbeault P, Almeras N, Tremblay A. Physical activity and low-fat diet: is it enough to maintain weight stability in the reduced-obese individual following weight loss by drug therapy and energy restriction? Obes Res. 1999 Jul;7(4):323-33. doi: 10.1002/j.1550-8528.1999.tb00415.x. PMID 10440588
- [Background] Doucet E, St-Pierre S, Almeras N, Imbeault P, Mauriege P, Pascot A, Despres JP, Tremblay A. Reduction of visceral adipose tissue during weight loss. Eur J Clin Nutr. 2002 Apr;56(4):297-304. doi: 10.1038/sj.ejcn.1601334. PMID 11965505
- [Background] Pare A, Dumont M, Lemieux I, Brochu M, Almeras N, Lemieux S, Prud'homme D, Despres JP. Is the relationship between adipose tissue and waist girth altered by weight loss in obese men? Obes Res. 2001 Sep;9(9):526-34. doi: 10.1038/oby.2001.69. PMID 11557833
- [Background] Krauss RM, Eckel RH, Howard B, Appel LJ, Daniels SR, Deckelbaum RJ, Erdman JW Jr, Kris-Etherton P, Goldberg IJ, Kotchen TA, Lichtenstein AH, Mitch WE, Mullis R, Robinson K, Wylie-Rosett J, St Jeor S, Suttie J, Tribble DL, Bazzarre TL. AHA Dietary Guidelines: revision 2000: A statement for healthcare professionals from the Nutrition Committee of the American Heart Association. Circulation. 2000 Oct 31;102(18):2284-99. doi: 10.1161/01.cir.102.18.2284. No abstract available. PMID 11056107
- [Background] Tremblay A, Despres JP, Maheux J, Pouliot MC, Nadeau A, Moorjani S, Lupien PJ, Bouchard C. Normalization of the metabolic profile in obese women by exercise and a low fat diet. Med Sci Sports Exerc. 1991 Dec;23(12):1326-31. PMID 1798373
- [Background] Burnham KP, Anderson DR. Model Selection and Inference. A Pratical Information-Theoretic Approach. Springer; 1998: Chapters 2.2, 2.4, pp43-48, pp51-54.